CLINICAL TRIAL: NCT05622877
Title: The Proteomic Study and Early Intervention Study of Carotid Unstable Plaque
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, jianwen guo, MD, professor, Guangzhou University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SZ2021ZZ3205
Record Dates: First submitted 2022-11-14; First posted 2022-11-21 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Protein; Disease; Carotid Artery Plaque; Traditional Chinese Medicine
Keywords: Traditional Chinese Medicine; proteomic study; carotid atherosclerosis plaques
MeSH Terms: conditions — Disease; Carotid Stenosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo Group (Placebo Comparator): Basic treatment according to the 2014 Chinese Guidelines for Secondary Prevention of Ischemic Stroke/Transient Ischemic Attack and placebo granules (6g/ bag, one bag each time, twice a day after meals);
  Interventions: Drug: placebo; Other: Basic treatment
- Qushi Formula Group (Experimental): Basic treatment according to the 2014 Chinese Guidelines for Secondary Prevention of Ischemic Stroke/Transient Ischemic Attack and Qushi Formula granules (6g/ bag, one bag each time, twice a day after meals);
  Interventions: Drug: Qushi Formula; Other: Basic treatment
- Zhu's Wenban Formula Group (Experimental): Basic treatment according to the 2014 Chinese Guidelines for Secondary Prevention of Ischemic Stroke/Transient Ischemic Attack and Zhu's Wenban Formula granules (6g/ bag, one bag each time, twice a day after meals);
  Interventions: Drug: Zhu's Wenban Formula; Other: Basic treatment

INTERVENTIONS:
Drug: Qushi Formula — Qushi Formula are decoction granules composed 8 traditional Chinese medicines, such as poria cocos, Macrocephalae Rhizoma, Polyporus, cassia twig, dried ginger and licorice, Etc.
  Arms: Qushi Formula Group
Drug: Zhu's Wenban Formula — Zhu's Wenban granules are decoction granules composed of leech, panax notoginseng, Atractylodes Lancea and rhizome
  Arms: Zhu's Wenban Formula Group
Drug: placebo — The placebo was composed of dextrin, powdered sugar, starch, and liquid caramel in the same color as the other two groups.
  Arms: Placebo Group
Other: Basic treatment — Basic diseases except hyperlipidemia were treated in accordance with the 2014 Chinese Guidelines for Secondary Prevention of Ischemic Stroke/Transient Ischemic Attack. Basic treatment includes conventional treatment such as comprehensive prevention and treatment (actively controlling basic diseases such as hypertension and diabetes and suggesting a good lifestyle), drug therapy (anti-inflammatory, lipid-regulating, anti-platelet aggregation, calcium channel blockers) and so on according to individual conditions of patients.

SUMMARY:
A study on the prediction model of carotid unstable plaque protein and its early intervention. Protein antibody chip was used to detect the remaining biological samples, and patients with carotid artery unstable plaque with stroke risk were selected for interventional clinical trials.

The selected patients were randomly divided into 3 groups, which were treated with Zhu's Wenban Formula (TCM compound granules), Qushi Formula (TCM compound granules) and placebo for 6 months, respectively. The size and number of carotid artery unstable plaques before and after 6 months were observed, and the occurrence of adverse reactions during the intervention period was observed.

ELIGIBILITY:
Inclusion Criteria:

* Wet syndrome scale assessment is consistent with wet syndrome diagnosis;
* Carotid color ultrasound indicated carotid artery unstable plaque.
* Protein chip analysis determined that the patients were at high risk of stroke
* Signing informed Consent

Exclusion Criteria:

* Carotid artery stenosis rate ≥50%;
* A definite or suspected diagnosis of vasculitis;
* Accompanied by infection, tumor, heart, liver and renal insufficiency (liver and
* kidney function more than twice the upper limit of normal value, cardiac function grade greater than or equal to 2);
* Patients with acute stroke or complicated with acute myocardial infarction and unstable angina pectoris;
* Pregnant or lactating women;
* A prior known allergy to the test drug or the test drug ingredient.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-05-31 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in carotid artery unstable plaque | 6 moths
  Changes in carotid IMT and the total volume and number of unstable plaques before and after 6 months of treatment

SECONDARY OUTCOMES:
Changes in blood lipids | 6 moths
  The changes of triglyceride, total cholesterol, low density lipoprotein and high density lipoprotein before and after 6 months of treatment;
Number of new cardiovascular events | 12 moths
  Number of cardiovascular and cerebrovascular events during 6 months of treatment and 6 months of follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Province Hospital of Tradtional Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided